CLINICAL TRIAL: NCT01519713
Title: Immunogenicity and Safety of a Single Dose of a Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (SP284) in Japanese Subjects
Brief Title: Study of a Single Dose of Meningococcal Polysaccharide Diphtheria Toxoid Conjugate Vaccine (SP284) in Japanese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA76 (SFY12080); U1111-1124-7479 (Other: WHO)
Record Dates: First submitted 2012-01-20; First posted 2012-01-27 (Estimated); Results first posted 2013-05-28 (Estimated); Last update posted 2013-05-28 (Estimated); Status verified 2013-05

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections
Keywords: Meningitis; Meningococcal Meningitis; Meningococcal Infections; Meningococcal conjugate Vaccine; Menactra®
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adults Study Group (Experimental): Participants will receive a single dose of Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate vaccine.
  Interventions: Biological: Meningococcal polysaccharide diphtheria toxoid conjugate
- Adolescents Study Group (Experimental): Participants will receive a single dose of Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate vaccine.
  Interventions: Biological: Meningococcal polysaccharide diphtheria toxoid conjugate
- Children Study Group (Experimental): Participants will receive a single dose of Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate vaccine.
  Interventions: Biological: Meningococcal polysaccharide diphtheria toxoid conjugate

INTERVENTIONS:
Biological: Meningococcal polysaccharide diphtheria toxoid conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®, SP284

SUMMARY:
This study is designed to assess the safety and immunogenicity of a single dose of Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (SP284) to support registration of the product in Japan.

Primary Objective:

* To describe the seroprotection rate [% of subjects with serum bactericidal assay using baby rabbit complement (SBA-BR) ≥1:128] to meningococcal antigens (serogroups A, C, Y and W-135) following vaccination with SP284 vaccine in subjects 2 through 55 years of age

Secondary Objectives:

* To describe the safety following receipt of SP284 vaccine in subjects 2 through 55 years of age
* To describe the immune responses to meningococcal antigens (serogroups A, C, Y and W-135) following vaccination with SP284 vaccine in subjects 2 through 55 years of age.

DETAILED DESCRIPTION:
All participants will receive a single injection of Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate vaccine on Day 0 and undergo immunogenicity assessment and safety monitoring post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 through 55 years on the day of inclusion
* For subjects ≥ 20 years of age: Informed consent form has been signed and dated by the subjects. For subjects 2 to 19 years of age: Informed consent form has been signed and dated by the parent(s) or other legal representative. Also subjects 7 to 11 years of age will provide assent and subjects 12 to 19 years of age will provide written assent form.
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman of childbearing potential, use of an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination.

Exclusion Criteria:

* Any acute and/or serious disease/illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* History of meningococcal diseases, confirmed either clinically, serologically, or microbiologically
* Known systemic hypersensitivity to any of the vaccine components, or history of a life threatening reaction to a vaccine containing the same substances of the study vaccine
* Known or suspected congenital or current/ previous acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroids therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial inclusion
* Planned participation in another clinical trial during the present trial period
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Receipt of any vaccine within the four weeks preceding the trial vaccination, except for influenza vaccination, which may be received at least two weeks before the study vaccine
* Planned receipt of any vaccine during the trial period
* Clinical or known serological evidence of systemic illness including hepatitis B, hepatitis C and/or human immunodeficiency virus (HIV) infection
* Ineligible according to the investigator's clinical judgment
* Known pregnancy, or suspected pregnancy or a positive (serum and/or urine) pregnancy test
* Currently breast feeding a child
* Known thrombocytopenia, contraindicating intramuscular (IM) vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Identified as employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family member (i.e., immediate, husband, wife and their children, adopted or natural) of the employees or the Investigator
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine
* History of Guillain-Barré Syndrome.

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Aventis K.K.
Locations (3):
- Japan (3):
  - Nagoya, Aichi-ken
  - Osaka, Osaka
  - Shinjuku, Tokyo

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 20 January through 25 February 2012 in 4 clinic sites in Japan.
Pre-assignment Details: A total of 200 subjects who met the inclusion, but no exclusion criteria were enrolled and vaccinated.
Groups:
- Adults Menactra® Vaccine Group: Participants aged 18 to 55 years received a single dose of Menactra® vaccine
- Adolescents Menactra® Vaccine Group: Participants aged 11 to 17 years received a single dose of Menactra® vaccine
- Children Menactra® Vaccine Group: Participants aged 2 to 10 years received a single dose of Menactra® vaccine
Period: Overall Study
Arm/Group | Adults Menactra® Vaccine Group | Adolescents Menactra® Vaccine Group | Children Menactra® Vaccine Group
Started | 194 | 2 | 4
Completed | 194 | 2 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adults Menactra® Vaccine Group | Adolescents Menactra® Vaccine Group | Children Menactra® Vaccine Group | Total
Number analyzed (Participants) | 194 | 2 | 4 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 4 | 6
  Between 18 and 65 years | 194 | 0 | 0 | 194
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 35.6 (11.2) | 11.0 (0.0) | 4.3 (2.6) | 34.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 0 | 2 | 99
  Male | 97 | 2 | 2 | 101
Region of Enrollment [Number; unit: Participants]
  Japan | 194 | 2 | 4 | 200

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serum Bovine Albumin Baby Rabbit (SBA-BR) Titers of >=1:128 Following Vaccination With One Dose of Menactra® Vaccine
Description: Functional antibody activity against meningococcal serogroups A, C, Y and W-135 antigens were determined by using a serum bovine assay using a baby rabbit complement (SBA-BR). Sero protection was defined as SBA-BR titer of ≥ 1:128.
Time Frame: 28 Days post-vaccination
Population: Functional antibody activity against meningococcal serogroups A, C, Y and W-135 antigens were determined in all enrolled and vaccinated participants, per-protocol population.
Measure: Number; unit: Participants
Arm/Group | Adults Menactra® Vaccine Group | Adolescents Menactra® Vaccine Group | Children Menactra® Vaccine Group
Number analyzed (Participants) | 194 | 2 | 4
Participants
  Serogroup A (N = 194, 2, 4) | 177 | 2 [0 to 0] | 4 [0 to 0]
  Serogroup C (N = 192, 2, 4) | 154 | 2 [0 to 0] | 4 [0 to 0]
  Serogroup Y (N = 192, 2, 4) | 180 | 2 [0 to 0] | 4 [0 to 0]
  Serogroup W-135 (N = 193, 2, 4) | 172 | 2 [0 to 0] | 4 [0 to 0]

2. Secondary Outcome: Number of Participants With Serum Bovine Albumin Baby Rabbit (SBA-BR) Titers of >=1:8 Following Vaccination With One Dose of Menactra® Vaccine
Description: Functional antibody activity against meningococcal serogroups A, C, Y and W-135 antigens were determined by using a serum bovine assay using a baby rabbit complement (SBA-BR).
Time Frame: 28 Days post-vaccination
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Adults Menactra® Vaccine Group | Adolescents Menactra® Vaccine Group | Children Menactra® Vaccine Group
Number analyzed (Participants) | 194 | 2 | 4
Participants
  Serogroup A (N = 194, 2, 4) | 180 | 2 [0 to 0] | 4 [0 to 0]
  Serogroup C (N = 192, 2, 4) | 167 | 2 [0 to 0] | 4 [0 to 0]
  Serogroup Y (N = 192, 2, 4) | 190 | 2 [0 to 0] | 4 [0 to 0]
  Serogroup W-135 (N = 193, 2, 4) | 186 | 2 [0 to 0] | 4 [0 to 0]

3. Secondary Outcome: Number of Participants With a 4-Fold Rise in Serum Bovine Albumin Baby Rabbit (SBA-BR) Titers on Day 28 From Day 0 Following Vaccination With One Dose of Menactra® Vaccine.
Description: as for outcome 2
Time Frame: 28 Days post-vaccination
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Adults Menactra® Vaccine Group | Adolescents Menactra® Vaccine Group | Children Menactra® Vaccine Group
Number analyzed (Participants) | 194 | 2 | 4
Participants
  Serogroup A (N = 193, 2, 4) | 150 | 2 [0 to 0] | 4 [0 to 0]
  Serogroup C (N = 191, 2, 4) | 151 | 2 [0 to 0] | 3 [0 to 0]
  Serogroup Y (N = 191, 2, 4) | 139 | 1 [0 to 0] | 4 [0 to 0]
  Serogroup W-135 (N = 192, 2, 4) | 169 | 2 [0 to 0] | 4 [0 to 0]

4. Secondary Outcome: Serum Bovine Albumin Baby Rabbit (SBA-BR) Geometric Mean Titers Following Vaccination With One Dose of Menactra® Vaccine
Description: as for outcome 2
Time Frame: Days 0 and 28 post-vaccination
Population: Geometric mean titers of antibodies against meningococcal serogroups A, C, Y and W-135 antigens were determined in all enrolled and vaccinated participants, per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Adults Menactra® Vaccine Group | Adolescents Menactra® Vaccine Group | Children Menactra® Vaccine Group
Number analyzed (Participants) | 194 | 2 | 4
Titers
  Serogroup A (Day 0; N = 193, 2, 4) | 26.0 [17.4 to 38.9] | 2.0 [NA to NA] — Data was not computable, variance was zero because all participants had the same value. | 2.0 [NA to NA] — Data was not computable, variance was zero because all participants had the same value.
  Serogroup A (Day 28; N = 194, 2, 4) | 1202.6 [876.2 to 1650.6] | 2896.3 [35.4 to 236766.0] | 16384.0 [1804.7 to 148741.4]
  Serogroup C (Day 0; N = 193, 2, 4) | 5.6 [4.2 to 7.4] | 2 [NA to NA] — Data was not computable, variance was zero because all participants had the same value. | 5.7 [0.2 to 154.7]
  Serogroup C (Day 28; N = 192, 2, 4) | 389.1 [274.4 to 551.8] | 2048.0 [0.0 to 91459214176.9] | 512.0 [208.0 to 1260.0]
  Serogroup Y (Day 0; N = 193, 2, 4) | 64.2 [45.1 to 91.5] | 181.0 [2.2 to 14797.9] | 107.6 [26.9 to 431.2]
  Serogroup Y (Day 28; N = 192, 2, 4) | 1244.4 [991.3 to 1562.2] | 724.1 [0.0 to 395556106.8] | 3444.3 [298.5 to 39740.1]
  Serogroup W-135 (Day 0; N = 193, 2, 4) | 12.8 [9.3 to 17.6] | 128.0 [0.0 to 855379.3] | 38.1 [1.4 to 1025.1]
  Serogroup W-135 (Day 28; N = 193, 2, 4) | 995.0 [737.9 to 1341.7] | 8192.0 [1.2 to 54744273.9] | 9742.0 [2431.7 to 39028.6]

5. Secondary Outcome: Serum Bovine Albumin Baby Rabbit (SBA-BR) Geometric Mean of Individual Titer Ratio Following Vaccination With One Dose of Menactra® Vaccine
Description: as for outcome 2
Time Frame: 28 Days post-vaccination
Population: Geometric mean titer ratios of antibodies against meningococcal serogroups A, C, Y and W-135 antigens were determined in all enrolled and vaccinated participants, per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Adults Menactra® Vaccine Group | Adolescents Menactra® Vaccine Group | Children Menactra® Vaccine Group
Number analyzed (Participants) | 194 | 2 | 4
Titers
  Serogroup A (N = 193, 2, 4) | 31.9 [21.7 to 46.8] | 724.1 [8.9 to 59191.5] | 4096.0 [451.2 to 37185.3]
  Serogroup C (N = 191, 2, 4) | 40.8 [28.3 to 58.9] | 512.0 [0.0 to 22864803544.2] | 53.8 [1.6 to 1838.6]
  Serogroup Y (N = 191, 2, 4) | 16.1 [11.6 to 22.2] | 4.0 [0.0 to 26730.6] | 32.0 [3.5 to 290.5]
  Serogroup W-135 (N = 192, 2, 4) | 53.6 [38.9 to 73.9] | 64.0 [NA to NA] — Data was not computable, variance was zero because all participants had the same value. | 215.3 [3.3 to 13841.7]

6. Secondary Outcome: Number of Participants Reporting at Least One Solicited Injection Site or Systemic Reactions Following Vaccination With One Dose of Menactra® Vaccine
Description: Solicited injection site reactions: Pain, Erythema and Swelling. Solicited systemic reactions: Fever (temperature), Headache, Malaise, and Myalgia.
  Grade 3 solicited reactions were defined as: Pain incapacitating (children) and prevents daily activities (adolescents and adults). Fever ≥ 39.0°C; Headache, Malaise and Myalgia, significant, prevents daily activities.
Time Frame: Day 0 up to Day 28 post-vaccination
Population: Solicited injection site and systemic reactions were assessed in all enrolled and vaccinated participants, Intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Adults Menactra® Vaccine Group | Adolescents Menactra® Vaccine Group | Children Menactra® Vaccine Group
Number analyzed (Participants) | 194 | 2 | 4
Participants
  Any injection site Pain | 60 | 0 [0 to 0] | 3 [0 to 0]
  Grade 3 injection site Pain | 0 | 0 [0 to 0] | 0 [0 to 0]
  Any injection site Erythema | 5 | 2 [0 to 0] | 3 [0 to 0]
  Grade 3 injection site Erythema | 0 | 1 [0 to 0] | 0 [0 to 0]
  Any injection site Swelling | 2 | 2 [0 to 0] | 3 [0 to 0]
  Grade 3 injection site Swelling | 0 | 0 [0 to 0] | 0 [0 to 0]
  Any Fever | 3 | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Fever | 0 | 0 [0 to 0] | 0 [0 to 0]
  Any Headache | 22 | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Headache | 0 | 0 [0 to 0] | 0 [0 to 0]
  Any Malaise | 30 | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Malaise | 3 | 0 [0 to 0] | 0 [0 to 0]
  Any Myalgia | 48 | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Myalgia | 1 | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected following vaccination on Day 0 up to Day 28 post-vaccination
Arm/Group | Adults Menactra® Vaccine Group | Adolescents Menactra® Vaccine Group | Children Menactra® Vaccine Group
Serious Adverse Events (participants affected / at risk) | 0/194 | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 63/194 | 2/2 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults Menactra® Vaccine Group (N=194) | Adolescents Menactra® Vaccine Group (N=2) | Children Menactra® Vaccine Group (N=4)
Injection site pain (General disorders) | 60 (60) | 0 (0) | 3 (3)
Injection site erythema (General disorders) | 5 (5) | 2 (2) | 3 (3)
Injection site swelling (General disorders) | 2 (2) | 2 (2) | 3 (3)
Malaise (General disorders) | 30 (30) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 48 (48) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 15 (17) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.